CLINICAL TRIAL: NCT05956041
Title: A Phase II Study of Pembrolizumab and Mogamulizumab in Advanced-stage, Relapsed/Refractory Cutaneous T-cell Lymphomas
Brief Title: Pembrolizumab and Mogamulizumab in Advanced-stage, Relapsed/Refractory Cutaneous T-cell Lymphomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2022.116; HUM00231051 (Other: University of Michigan); HCRN (Other: LYM21-546)
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous T Cell Lymphoma; Fungoides Mycosis Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — pembrolizumab; mogamulizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental): Pembrolizumab 400mg via IV over 30 minutes on Day 1 of each cycle (6 weeks) Mogamulizumab 1mg/kg via IV over a least 60 minutes Cycle 1: Days 1, 8, 15, and 22 Cycle 2+: Days 1, 15, and 29 Each cycle lasts 6 weeks with a maximum of 18 cycles If a subject achieves a complete response (CR) after 3 months of study treatment (2 cycles), they will continue study therapy for an additional 6 months (4 cycles). If a confirmed and persistent CR they may discontinue study treatment and enter an observation period. Subjects who progress during the observation period may be eligible for up to an additional 12 cycles of pembrolizumab and mogamulizumab
  Interventions: Drug: Pembrolizumab; Drug: Mogamulizumab

INTERVENTIONS:
Drug: Pembrolizumab — 400mg Intravenously
  Other Names: Keytruda
Drug: Mogamulizumab — 1mg/kg Intravenously
  Other Names: Poteligeo

SUMMARY:
This is an open-label, single-arm, multicenter, phase II study combining pembrolizumab and mogamulizumab in patients with advanced-stage, relapsed or refractory CTCL Each cycle will equal 6 weeks. Pembrolizumab will be administered on Day 1 of each cycle. Mogamulizumab will be administered on Day 1, 8, 15, and 22 of Cycle 1. For Cycle 2 and subsequent cycles, mogamulizumab will be administered on Day 1, 15 and 29 of each cycle. Subjects will undergo a response assessment prior to Cycle 3 and every 2 cycles thereafter.

Subjects will continue study treatment until documented progression, unacceptable toxicity, or any other condition for discontinuation is met in protocol. A maximum of 2 years of study treatment may be administered. If a subject achieves a complete response (CR) per mSWAT criteria after 3 months of study treatment (2 cycles), they will continue study therapy for an additional 6 months (4 cycles). If a confirmed and persistent CR is met, they may discontinue study treatment and enter an observation period in protocol. Repeat disease evaluation is required prior to study therapy discontinuation. Subjects who progress during the observation period may be eligible for up to an additional 9 cycles (1 year) of pembrolizumab and mogamulizumab.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of ≤ 1 within 7 days prior to Cycle 1 Day 1 treatment.
* Histological confirmation of cutaneous T-cell lymphoma (Mycosis Fungoides/Sezary Syndrome) with Stage IIB-IVB disease (TNMB Classification).
* Measurable disease according to Modified Severity Weighted Assessment Tool (mSWAT) within 30 days prior to treatment.
* Patients must have measurable, unirradiated disease. Prior disease radiation, if greater than 7 days prior to C1D1, is acceptable (see protocol). However, patient must have measurable disease that has not been radiated.
* Patients must have failed at least one prior line of systemic therapy. This includes ECP. Prior cancer treatment must be completed at least 28 days prior to Cycle 1 Day 1(C1D1) and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤ grade 1 or baseline.
* Archival tissue is required and will be identified at screening and shipped prior to C1D1 (10-15 unstained slides; obtained within 90 days of registration). Subjects that do not have archival tissue will be required to undergo a skin biopsy.
* Systemic steroids at a dose less than the equivalent of 10 mg/day of prednisone and inhaled, nasal, and topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease are permitted. Treatment with a short course of steroids (< 5 days) up to 7 days prior to study registration is permitted.
* Demonstrate adequate organ function as defined below. All screening labs to be obtained within 28 days prior to Cycle 1 Day 1.

  * Hematological
  * Absolute Neutrophil Count (ANC) ≥ 500/µL
  * Hemoglobin (Hgb) ≥ 8 g/dL
  * Platelet Count ≥ 25 000/µL
  * Renal

    ---Creatinine OR Measured or calculated creatinine clearance1 ≤ 1.5 × ULN OR

    ≥ 30 mL/min for participant with creatinine levels > 1.5 × institutional ULN
  * Hepatic
  * Bilirubin ≤ 1.5 ×ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases)
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases)
  * Coagulation ---International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Females of childbearing potential must have a negative serum pregnancy test within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. See protocol for definition of childbearing potential.
* Females of childbearing potential must be willing to abstain from heterosexual intercourse or to use an effective method(s) of contraception as outlined in protocol. Males must be willing to abstain from heterosexual intercourse or to use an effective method(s) of contraception as outlined in protocol.
* Subjects with CNS disease are eligible so long as they meet all other eligibility criteria.
* Patients must have a life expectancy of at least 6 months.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Patients with a known history of Human Immunodeficiency Virus (HIV) infection are excluded. NOTE: No HIV testing is required unless mandated by local health authority.
* Patients with concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection. NOTE: Hepatitis B and C screening tests are not required unless: (1) Known history of HBV and HCV infection or (2) As mandated by local health authority.
* Patients previously treated with checkpoint blockade, including pembrolizumab, or mogamulizumab, are excluded.
* Patients who have received disease radiation therapy within 7 days of C1D1.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to Cycle 1 Day 1. Systemic steroids at a dose less than the equivalent of 10 mg/day of prednisone and inhaled, nasal, and topical steroids are permitted as detailed in protocol.
* Has active or prior autoimmune disease or inflammatory disorders that have required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs) with teh exception of vitiligo or alopecia. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Known additional malignancy that is progressing or has required active treatment within the past 2 years. NOTE: patients with non-melanoma skin cancers and in situ cancers that do not require systemic therapies are eligible.
* Active infection requiring systemic therapy.
* Prior allogeneic stem cell transplant or allogeneic cellular therapies, recent immunosuppressive therapies (for any reason).
* Prior solid organ transplant.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab or mogamulizumab and/or any of their excipients.
* Treatment with any investigational drug or investigation device within 30 days prior to registration.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines and mRNA or inactivated COVID-19 vaccine is allowed.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | 6 months
  Complete response (CR) rate at 6 months. CR is defined as percentage of patients who have a best response of CR at 6 months using mSWAT response criteria.

SECONDARY OUTCOMES:
Best overall Response (BOR) | 2 years
  Best overall response (BOR) is defined as the best response recorded from the start of the treatment until progression/recurrence using mSWAT response criteria
Duration of response (DOR) | 2 years
  Duration of response (DOR) is defined as time from first observed response (CR or PR) to date of progression (PD) or death, whichever occurs first using mSWAT response criteria
Time to next treatment (TTNT) | 2 years
  Time to next treatment (TTNT) is defined as time from Cycle 1 Day 1 to initiation of alternative systemic, antineoplastic therapy
Assess Adverse Events | 2 years
  Safety will be determined based on the frequency and severity of adverse events according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5. Specifically, grade 3-4 adverse events related to study treatment affecting 10% or more of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Wilcox, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No